CLINICAL TRIAL: NCT00285922
Title: Comparison of Estimated Body Surface Potential Mapping With Standard Electrocardiography in Patients Presenting to the Emergency Department With Chest Pain
Brief Title: Novel Method to Diagnose Acute Myocardial Ischemia
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Other Study IDs: RO1 HL69758-10
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-02-02 (Estimated); Status verified 2005-07

CONDITIONS: Myocardial Infarction; Angina, Unstable; Myocardial Ischemia; Coronary Disease
Keywords: myocardial infarction; electrocardiography; myocardial ischemia; emergency medicine; monitoring, physiologic
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aim of this study is to improve the detection of heart attack in people who come to a hospital emergency room (ER) with cardiac symptoms. We are testing a novel technology that calculates the heart's electrical activity at points all around the upper body torso and develops a map showing areas indicating heart attack. Our hypothesis is that this new body mapping technique will be better than the standard electrocardiogram (ECG) in detecting heart attack.

DETAILED DESCRIPTION:
The overall aims of the proposed research are (1) to improve the ECG diagnosis of patients who present to the ER with heart attack and (2) to improve the monitoring of recurrent heart attack in these patients while they are being treated in the hospital. The proposed research will test a promising new technique, termed estimated body surface potential mapping. This novel method involves estimating ECG information across the entire upper body from 10 electrodes placed in strategic positions.

In patients who come to the ER complaining of chest pain, shortness of breath or some other symptom of a heart attack, we will: (1) record continuous, 24 hour, standard ECGs (usual, current method used) and at the same time (2)record continuous 24 hour experimental recordings from which a body surface map will be calculated. Two experts who do not know whether the patient actually had a heart attack or not will analyze these 2 methods for signs of heart attack. We expect that more correct diagnoses will happen with the new experimental body mapping technique. The correct diagnosis will be based upon a blood test which is considered the best test to prove there is heart damage. The blood test does not become abnormal until hours after the attack, however, so the ECG diagnosis must be made and treatment initiated before results of the blood test are available.

If the expected diagnostic improvements are confirmed in this study, the long term benefit would be more accurate ER decision-making of patients with heart attack and more timely treatment. The benefits of more timely and definitive treatment would be an improvement in long-term survival, functional status, and quality of life in patients treated for heart attack.

We plan to enroll 1,320 patients who present to the ER at the University of California, San Franicsco to participate in the study. We will follow these patients for a year following their ER visit to determine whether they survived and which ECG method predicted death more accurately.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who present to the UCSF emergency room between 7 am and 7 pm, Monday through Friday, who have symptoms of myocardial infarction.

Exclusion Criteria:

* Patients with left bundle branch block or ventricular pacemaker rhythm

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320
Dates: Start 2001-08; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Drew, PhD, Principal Investigator — University of California, San Francisco; Robert M Lux, PhD, Study Director — University of Utah, Salt Lake
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Lux R, Bilbao M, Pelter M, Fleischmann K, Zegre J, Schindler D, Drew B. Optimal leads, estimation, and continuous monitoring improve detection of acute MI and transient ischemia. J Electrocardiol. 2004;37 Suppl:240-3. doi: 10.1016/j.jelectrocard.2004.08.064. No abstract available. PMID 15534848
- See also: Faculty profile — http://nurseweb.ucsf.edu/www/ffdrew.htm//